CLINICAL TRIAL: NCT03034421
Title: Prevention of Pneumothorax Following Endoscopic Valve Therapy in Patients With Severe Emphysema
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficult patient recruitment
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Felix JF Herth, Prof. Dr. med., Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Protocol G1.1 - 17.04.2016
Record Dates: First submitted 2016-09-16; First posted 2017-01-27 (Estimated); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Pneumothorax
MeSH Terms: conditions — Pneumothorax | interventions — Bed Rest

ARMS (2):
- Modified medical care (Active Comparator): Patients will undergo 48-hours bed rest after endoscopic valve implantation.
  Interventions: Behavioral: Bed rest
- Standard medical care (No Intervention): Patients will be treated with standard medical care without restriction to bed rest after endoscopic valve implantation.

INTERVENTIONS:
Behavioral: Bed rest — Patients will undergo bed rest for 48 hours following endoscopic valve implantation.
  Arms: Modified medical care

SUMMARY:
Endoscopic valve therapy is an effective therapy for patients with severe emphysema and low interlobar collateral ventilation. Although, valve therapy is a minimal-invasive treatment approach, it is associated with complications the most common of which is pneumothorax with a rate of 18-25%. Modifying post-operative medical care including bed rest for 48 hours after valve implantation may reduce the risk of post-interventional pneumothorax.

DETAILED DESCRIPTION:
Patient enrolment and data acquisition is to be carried out on a prospective basis. It is planned to enrol a total of 130 patients with advanced emphysema and low collateral ventilation. Patients will be randomly assigned in a 1:1 ratio to receive modified medical care including a 48 bed rest or standard medical care following valve implantation. All patients will undergo treatment at one study centre in Heidelberg.

ELIGIBILITY:
Inclusion Criteria:

* FEV1 < 50%, RV>150%, TLC>100%
* emphysema confirmed by computed tomography
* pO2 >60 mmHg (with supplemental oxygen), pCO2 < 55 mmHg (room condition)
* no significant collateral ventilation (assessed by fissure analysis and/or catheter-based measurement)
* no COPD exacerbation within the past 8 weeks
* daily use of < 20 mg Prednisolon
* non-smoking for a minimum of 4 months prior to consent
* Patient has provided written informed consent

Exclusion Criteria:

* BMI < 18 kg/m²
* clinically relevant bronchiectasis
* failed cardiac clearance: defined as myocardial infarction within last 6 weeks, decompensation of heart failure
* Prior lung resection (e.g. lobectomy)

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-09; Primary Completion 2018-08-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Advent of pneumothorax within 90 days following valve implantation | 90 days following valve implantation
  Incidence of pneumothorax that is confirmed by radiological procedures within 90 days after implantation of valves.

SECONDARY OUTCOMES:
Lung function before and after valve therapy | 30 and 90 days following valve implantation
  Lung function parameters (VC [L], FEV1 [L], RV [L], TLC [L] will be assessed 30 and 90 days following valve implantation.
Excercise capacity before and after valve therapy | 30 and 90 days following valve implantation
  6-minute-walk test (m) will be assessed 30 and 90 days following valve implantation.
Dyspnoe score before and after valve therapy | 30 and 90 days following valve implantation
  Dyspnoe score (mMRC) will be assessed 30 and 90 days following valve implantation.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Gompelmann, MD, Principal Investigator — Thoraxklinik at University of Heidelberg
Locations (1):
- Thoraxklinik Heidelberg, Heidelberg, Germany